CLINICAL TRIAL: NCT03458910
Title: Why Does Heart Rate Variability Matter for Emotion Regulation
Brief Title: Heart Rate Variability and Emotion Regulation
Acronym: HRV-ER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 increased risk of participation
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Mara Mather, Professor of Gerontology and Psychology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UP-17-00219
Record Dates: First submitted 2018-02-13; First posted 2018-03-08 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Heart Rate Variability
Keywords: heart rate variability, HRV

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the HRV-increase group or the HRV-decrease group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV-increase group (Experimental): Half of the participants will be randomly assigned to this group who will undergo daily practice to increase their heart rate variability (HRV).
  Interventions: Behavioral: HRV training
- HRV-decrease group (Experimental): Half of the participants will be randomly assigned to this group who will undergo daily practice to decrease their HRV and heart rate.
  Interventions: Behavioral: HRV training

INTERVENTIONS:
Behavioral: HRV training — Participants will be asked to undergo daily practice to regulate (either increase or decrease) HRV for 5 weeks.

SUMMARY:
Previous research suggests that heart rate variability (HRV) biofeedback aimed at increasing HRV can reduce anxiety and stress. However, some mental quiescence practices that reduce HRV during the practice sessions also lead to positive emotional outcomes. Thus, it is not obvious that the benefits of HRV-biofeedback accrue due to increasing HRV during the session. An alternative possibility is that the benefits arise from engaging prefrontal control over heart rate. In this study, the investigators will test two possible mechanisms of the effects of HRV on emotional health by comparing two groups. In one group, participants will be asked to engage in daily training to decrease HRV using the HRV biofeedback device. In the other group, participants will be asked to engage in daily training to increase HRV using the HRV biofeedback device. This will allow analyses to pit two possible mechanisms against each other:

1. Mechanism 1: engaging prefrontal control over heart rate is the critical factor that allows HRV biofeedback to help improve well-being. In this case, well-being should increase over time in both groups, as both training should engage prefrontal cortex to implement self-directed control over heart rate. Strengthening prefrontal control mechanisms may help improve emotion regulation in everyday life.
2. Mechanism 2: increased HRV during the training sessions leads to greater functional connectivity among brain regions associated with emotion regulation during the high HRV state. In this case, improved well-being would be specifically associated with having time each day during which there were very high HRV states, and so improved well-being should be seen only in the group in which participants get biofeedback to increase HRV.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Aged between 18-35 for the younger group and aged between 55-80 for the older group
* Scores on TELE indicate no current dementia
* Normal or corrected-to-normal vision and hearing
* People taking antidepressant, anti-anxiety medication and/or attending psychotherapy only if the treatment had been ongoing and unchanged for at least three months

Exclusion Criteria:

* Have a disorder that would impede performing the HRV biofeedback procedures (i.e., abnormal cardiac rhythm, heart disease including coronary artery disease, angina, and arrhythmia, cardiac pacemaker, stroke, panic attack, cognitive impairment).
* Current practice of any relaxation, biofeedback, or breathing technique.
* Currently taking any psychoactive drugs other than antidepressants or anti-anxiety medications
* No trips that would lead them to miss any of the weekly meetings
* Currently nursing, pregnant, or intend to become pregnant
* Have metals in their body, as this is a scanning requirement
* Have any conditions listed in the MRI Screening form (see below)

MRI screening

* Cardiac pacemaker
* Implanted cardiac defibrillator
* Aneurysm clip or brain clip
* Carotid artery vascular clamp
* Neurostimulator
* Insulin or infusion pump
* Spinal fusion stimulator
* Cochlear, otologic, ear tubes or ear implant
* Prosthesis (eye/orbital, penile, etc.)
* Implant held in place by a magnet
* Heart valve prosthesis
* Artificial limb or joint
* Other implants in body or head
* Electrodes (on body, head or brain)
* Intravascular stents, filters, or
* Shunt (spinal or intraventricular)
* Vascular access port or catheters
* IUD or diaphragm
* Transdermal delivery system or other types of foil
* patches (e.g. Nitro, Nicotine, Birth control, etc.)
* Shrapnel, buckshot, or bullets
* Tattooed eyeliner or eyebrows
* Body piercing(s)
* Metal fragments (eye, head, ear, skin)
* Internal pacing wires
* Aortic clips
* Metal or wire mesh implants
* Wire sutures or surgical staples
* Harrington rods (spine)
* Bone/joint pin, screw, nail, wire, plate
* Wig, toupee, or hair implants
* Asthma or breathing disorders
* Seizures or motion disorders
* Hospitalization for mental or neurological illness
* Head Trauma
* Migraine Headache
* Panic attack
* Stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Mather, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Min J, Rouanet J, Martini AC, Nashiro K, Yoo HJ, Porat S, Cho C, Wan J, Cole SW, Head E, Nation DA, Thayer JF, Mather M. Modulating heart rate oscillation affects plasma amyloid beta and tau levels in younger and older adults. Sci Rep. 2023 Mar 9;13(1):3967. doi: 10.1038/s41598-023-30167-0. PMID 36894565
- [Derived] Cho C, Yoo HJ, Min J, Nashiro K, Thayer JF, Lehrer PM, Mather M. Changes in Medial Prefrontal Cortex Mediate Effects of Heart Rate Variability Biofeedback on Positive Emotional Memory Biases. Appl Psychophysiol Biofeedback. 2023 Jun;48(2):135-147. doi: 10.1007/s10484-023-09579-1. Epub 2023 Jan 20. PMID 36658380

RESULTS

PARTICIPANT FLOW:
Groups:
- Younger HRV-increase Group: Participants in this group were between the ages of 18 and 35.
  Half of the younger participants were randomly assigned to this group and underwent daily practice to increase their heart rate variability (HRV) for 5 weeks.
- Younger HRV-decrease Group: Participants in this group were between the ages of 18 and 35.
  Half of the younger participants were randomly assigned to this group and underwent daily practice to decrease their heart rate variability (HRV) for 5 weeks.
- Older HRV-increase Group: Participants in this group were between the ages of 55 and 80.
  Half of the older participants were randomly assigned to this group and underwent daily practice to increase their heart rate variability (HRV) for 5 weeks.
- Older HRV-decrease Group: Participants in this group were between the ages of 55 and 80.
  Half of the older participants were randomly assigned to this group and underwent daily practice to decrease their heart rate variability (HRV) for 5 weeks.
Period: Overall Study
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group | Older HRV-increase Group | Older HRV-decrease Group
Started | 63 | 58 | 37 | 35
Completed | 56 | 50 | 28 | 28
Not Completed | 7 | 8 | 9 | 7
Not completed — Withdrawal by Subject | 7 | 8 | 6 | 4
Not completed — Study halted due to risk of catching COVID-19 | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group | Older HRV-increase Group | Older HRV-decrease Group | Total
Number analyzed (Participants) | 63 | 58 | 37 | 35 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 4 | 0 | 0 | 10
  Between 18 and 65 years | 57 | 54 | 21 | 14 | 146
  >=65 years | 0 | 0 | 16 | 21 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.71 (2.47) | 22.66 (3.17) | 65.03 (8.29) | 65.66 (5.88) | 38.68 (21.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 24 | 21 | 105
  Male | 32 | 29 | 13 | 14 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 3 | 12
  Not Hispanic or Latino | 55 | 48 | 35 | 31 | 169
  Unknown or Not Reported | 6 | 5 | 0 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 43 | 38 | 5 | 6 | 92
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 12 | 2 | 18
  White | 9 | 13 | 18 | 25 | 65
  More than one race | 2 | 2 | 2 | 1 | 7
  Unknown or Not Reported | 5 | 5 | 0 | 1 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 58 | 37 | 35 | 193

OUTCOME MEASURES:

1. Primary Outcome: mPFC-right Amygdala Resting-state Functional Connectivity for Younger Adults (ANOVA)
Description: The strength of resting-state functional connectivity was measured by correlation coefficients. Values represent the correlation of BOLD time-series between mPFC and the right amygdala. Higher values indicate greater connectivity.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: Population analyzed was composed by all randomization subjects who completed pre- and post-intervention assessments and whose data quality was sufficient for data analysis.
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 49 | 47
correlation coefficients
  Time 1 | 0.104 (0.105) | 0.086 (0.015)
  Time 2 | 0.116 (0.015) | 0.090 (0.015)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; A 2 (time: pre, post) X 2 (condition: HRV-increase, HRV-decrease) ANOVA was performed; Test type: Superiority; p = 0.782, ANOVA

2. Primary Outcome: mPFC-right Amygdala Resting-state Functional Connectivity for Older Adults (ANOVA)
Description: as for outcome 1
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 26 | 25
correlation coefficients
  Time 1 | 0.109 (0.045) | 0.140 (0.046)
  Time 2 | 0.125 (0.046) | 0.095 (0.047)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; A 2 (time: pre, post) X 2 (condition: HRV-increase, HRV-decrease) ANOVA was performed; Test type: Superiority; p = 0.480, ANOVA

3. Primary Outcome: mPFC-right Amygdala Resting-state Functional Connectivity for Younger Adults (Post-Pre)
Description: The strength of resting-state functional connectivity between mPFC and the right amygdala was measured by correlation coefficients. The difference in functional connectivity between the two time points (Time 2 - Time 1) was calculated. Higher values indicate greater connectivity at Time 2 than Time 1 (or post- than pre-intervention).
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 49 | 47
correlation coefficients | 0.011 (0.022) | -0.016 (0.024)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; An independent t-test was performed to compare the two groups; Test type: Superiority; p = 0.410, t-test, 2 sided

4. Primary Outcome: mPFC-right Amygdala Resting-state Functional Connectivity for Older Adults (Post-Pre)
Description: as for outcome 3
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 26 | 25
correlation coefficients | 0.016 (0.072) | -0.045 (0.046)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; An independent t-test was performed to compare the two groups; Test type: Superiority; p = 0.480, t-test, 2 sided

5. Secondary Outcome: Emotion Regulation in Younger Adults (Behavior)
Description: Emotional intensity ratings, which participants reported during the emotion regulation task inside MRI scanner before and after intervention. The ratings ranged from 1 through 4, and 4 represents strongest intensity.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 44 | 39
score on a scale
  Time 1: down-regulation | 1.841 (0.080) | 1.822 (0.085)
  Time 1: viewing | 2.073 (0.084) | 2.309 (0.089)
  Time 1: up-regulation | 3.141 (0.072) | 3.271 (0.076)
  Time 2: down-regulation | 1.861 (0.075) | 1.959 (0.080)
  Time 2: viewing | 1.964 (0.078) | 2.427 (0.083)
  Time 2: up-regulation | 3.269 (0.070) | 3.395 (0.074)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; time x condition x regulation goal interaction in behavioral emotional intensity rating for younger adults; Test type: Superiority; p = 0.170, ANOVA

6. Secondary Outcome: Emotion Regulation in Older Adults (Behavior)
Description: as for outcome 5
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 18 | 19
score on a scale
  Time 1: down-regulation | 2.059 (0.085) | 1.973 (0.119)
  Time 1: viewing | 2.586 (0.096) | 2.511 (0.134)
  Time 1: up-regulation | 3.117 (0.087) | 3.022 (0.121)
  Time 2: down-regulation | 2.115 (0.087) | 2.061 (0.122)
  Time 2: viewing | 2.668 (0.116) | 2.695 (0.162)
  Time 2: up-regulation | 3.279 (0.069) | 3.155 (0.097)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; time x condition x regulation goal interaction in behavioral emotional intensity rating for older adults; Test type: Superiority; p = 0.478, ANOVA

7. Secondary Outcome: Left Amygdala BOLD Activity During Emotion Regulation in Younger Adults
Description: We measured percent changes (%) in BOLD activity in the left amygdala region during emotion down-regulation, viewing, and up-regulation before and after intervention. The viewing condition was used as a baseline during the task. The change is represented by %.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent changes (%) in BOLD signal
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 45 | 39
Percent changes (%) in BOLD signal
  Time 1: down-regulation | 0.032 (0.022) | 0.024 (0.023)
  Time 1: viewing | 0.029 (0.023) | 0.048 (0.035)
  Time 1: up-regulation | 0.107 (0.026) | 0.095 (0.028)
  Time 2: down-regulation | 0.027 (0.021) | 0.021 (0.022)
  Time 2: viewing | 0.018 (0.019) | -0.020 (0.021)
  Time 2: up-regulation | 0.121 (0.027) | 0.074 (0.029)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; time x condition x regulation goal (2 x 2 x 3) interaction effect in the left amygdala for younger adults; Test type: Superiority; p = 0.441, ANOVA

8. Secondary Outcome: Left Amygdala BOLD Activity During Emotion Regulation in Older Adults
Description: as for outcome 7
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent changes (%) in BOLD signal
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 21 | 20
Percent changes (%) in BOLD signal
  Time 1: down-regulation | -0.069 (0.041) | -0.028 (0.043)
  Time 1: viewing | -0.092 (0.039) | -0.006 (0.040)
  Time 1: up-regulation | -0.043 (0.052) | 0.067 (0.053)
  Time 2: down-regulation | -0.068 (0.037) | -0.035 (0.038)
  Time 2: viewing | -0.004 (0.030) | -0.013 (0.031)
  Time 2: up-regulation | -0.013 (0.031) | 0.036 (0.032)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; time x condition x regulation goal (2 x 2 x 3) interaction effect in the left amygdala for older adults; Test type: Superiority; p = 0.621, ANOVA

9. Secondary Outcome: Right Amygdala BOLD Activity During Emotion Regulation in Younger Adults
Description: We measured percent changes (%) in BOLD activity in the right amygdala region during emotion down-regulation, viewing, and up-regulation before and after intervention. The viewing condition was used as a baseline during the task. The change is represented by %.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent changes (%) in BOLD signal
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 45 | 39
Percent changes (%) in BOLD signal
  Time 1: down-regulation | 0.019 (0.021) | 0.018 (0.023)
  Time 1: viewing | 0.032 (0.021) | 0.039 (0.022)
  Time 1: up-regulation | 0.054 (0.024) | 0.074 (0.025)
  Time 2: down-regulation | 0.076 (0.026) | 0.017 (0.028)
  Time 2: viewing | 0.073 (0.027) | -0.003 (0.029)
  Time 2: up-regulation | 0.106 (0.025) | 0.068 (0.027)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; time x condition x regulation goal (2 x 2 x 3) interaction effect in the right amygdala activity for younger adults; Test type: Superiority; p = 0.190, ANOVA

10. Secondary Outcome: Right Amygdala BOLD Activity During Emotion Regulation in Older Adults
Description: as for outcome 9
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent changes (%) in BOLD signal
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 21 | 20
Percent changes (%) in BOLD signal
  Time 1: down-regulation | -0.058 (0.052) | -0.014 (0.053)
  Time 1: viewing | 0.005 (0.029) | -0.027 (0.030)
  Time 1: up-regulation | 0.041 (0.045) | 0.062 (0.047)
  Time 2: down-regulation | -0.038 (0.031) | -0.004 (0.032)
  Time 2: viewing | -0.005 (0.027) | 0.001 (0.027)
  Time 2: up-regulation | 0.006 (0.038) | 0.024 (0.039)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; time x condition x regulation goal (2 x 2 x 3) interaction effect in the right amygdala activity for older adults; Test type: Superiority; p = 0.864, ANOVA

11. Secondary Outcome: Decision-making for Younger Adults at Post Intervention (Behavior)
Description: The decision-making ability was measured by multiple-choice responses during a computer-based task.
  Median percentage of acceptance of unfair offers and fair offers were calculated.
  A higher percentage of accepted both unfair and fair offers points toward more rational decision-making and likely better emotion regulation.
  This task was administered only at post-intervention (but not pre-intervention).
Time Frame: one time point: at study completion, which is the end of 5-week training
Population: Population analyzed was composed by all randomization subjects who completed the decision making task, who were unfamiliar with the task and whose data quality was sufficient for data analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of offers
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 35 | 33
percentage of offers
  percentage of acceptance of fair offers | 100 [100 to 100] | 100 [100 to 100]
  percentage of acceptance of unfair offers | 33.33 [5.56 to 72.22] | 33.33 [5.72 to 80.21]
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Comparing acceptance rate of fair offers; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Comparing acceptance rate of unfair offers; Test type: Superiority; p = 0.716, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Decision-making for Younger Adults (fMRI)
Description: We measured percent changes (%) in BOLD activity in the dorsal anterior cingulate cortex and anterior insula during a computer-based decision-making task. Higher values indicate greater activity.
Time Frame: one time point: at study completion, which is the end of 5-week training
Population: Population analyzed was composed by all randomization subjects who completed the decision making task, whose data quality was sufficient for data analysis and who were unfamiliar with the task.
Measure: Mean (Standard Error); unit: Percent changes (%) in BOLD signal
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 31 | 30
Percent changes (%) in BOLD signal
  Dorsal anterior cingulate cortex activation | 0.1073 (0.0221) | 0.0177 (0.0278)
  Anterior insula activation | 0.0740 (0.0214) | 0.0135 (0.0229)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; An independent t-test was performed to compare the two groups for dorsal anterior cingulate cortex activation; Test type: Superiority; p = 0.014, t-test, 2 sided
Statistical Analysis 2: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; An independent t-test was performed to compare the two groups for anterior insula activation; Test type: Superiority; p = 0.059, t-test, 2 sided

13. Secondary Outcome: Mood for Younger Adults
Description: Emotional well-being measured by the Profile of Mood States (POMS) for younger adults.
  The POMS consists of 40 items that are rated on a 5-point scale ranging from "0=not at all" to "4=extremely. Total Mood Disturbance (TMD) was calculated by summing the totals for the negative items and then subtracting the totals for the positive items. A constant (i.e., 100) was added to the TMD formula in order to eliminate negative scores. Higher scores indicate more negative mood states. The scores range from 56 and 216.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 53 | 50
score on a scale
  Time 1 | 92.604 (14.270) | 93.560 (18.307)
  Time 2 | 89.726 (18.710) | 86.540 (18.967)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = .144, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores
Statistical Analysis 2: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.653, Mixed Models Analysis — Linear mixed effects model with random factors (intercepts) for participants; F- and p-values determined using Satterthwaite's method

14. Secondary Outcome: Mood for Older Adults
Description: Emotional well-being measured by the Profile of Mood States (POMS) for older adults.
  The POMS consists of 40 items that are rated on a 5-point scale ranging from "0=not at all" to "4=extremely. Total Mood Disturbance (TMD) was calculated by summing the totals for the negative items and then subtracting the totals for the positive items. A constant (i.e., 100) was added to the TMD formula in order to eliminate negative scores. Higher scores indicate more negative mood states. The scores range from 56 and 216.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 27 | 28
score on a scale
  Time 1 | 87.167 (17.435) | 90.250 (17.037)
  Time 2 | 79.852 (12.440) | 87.536 (18.339)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = .288, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores
Statistical Analysis 2: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.191, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 2]; p-value reflects effect of interest, a time x condition interaction on scores

15. Secondary Outcome: Depression for Younger Adults
Description: Emotional well-being measured by the Center for Epidemiological Studies Depression Scale (CES-D) for younger adults.
  The CES-D consists of 20 items that are rated on a scale of 0 to 3 (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Possible range of scores is 0 to 60, with the higher scores indicating more depressive symptoms.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 55 | 49
score on a scale
  Time 1 | 16.164 (8.046) | 14.571 (9.372)
  Time 2 | 13.218 (8.774) | 11.837 (8.880)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.894, ANOVA
Statistical Analysis 2: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.425, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 2]; p-value reflects effect of interest, a time x condition interaction on scores

16. Secondary Outcome: Depression for Older Adults
Description: Emotional well-being measured by the Center for Epidemiological Studies Depression Scale (CES-D) for older adults.
  The CES-D consists of 20 items that are rated on a scale of 0 to 3 (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Possible range of scores is 0 to 60, with the higher scores indicating more depressive symptoms.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 27 | 28
score on a scale
  Time 1 | 8.852 (7.383) | 14.143 (9.816)
  Time 2 | 6.481 (4.839) | 11.964 (8.963)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.916, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores
Statistical Analysis 2: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.235, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 2]; p-value reflects effect of interest, a time x condition interaction on scores

17. Secondary Outcome: State Anxiety for Younger Adults
Description: Emotional well-being measured by the State Anxiety Inventory (SAI) for younger adults.
  The SAI consists of 20 items that are rated on a 4-point scale as follows: 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Scores range from 20 to 80, with higher scores indicating greater state anxiety.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 53 | 49
score on a scale
  Time 1 | 38.566 (10.233) | 38.122 (11.245)
  Time 2 | 37.972 (10.511) | 36.347 (11.816)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.462, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores
Statistical Analysis 2: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.468, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 2]; p-value reflects effect of interest, a time x condition interaction on scores

18. Secondary Outcome: State Anxiety for Older Adults
Description: Emotional well-being measured by the State Anxiety Inventory (SAI) for older adults.
  The SAI consists of 20 items that are rated on a 4-point scale as follows: 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Scores range from 20 to 80, with higher scores indicating greater state anxiety.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 28 | 27
score on a scale
  Time 1 | 31.786 (8.741) | 33.889 (11.078)
  Time 2 | 30.143 (7.966) | 33.963 (10.082)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.481, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores
Statistical Analysis 2: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.159, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 2]; p-value reflects effect of interest, a time x condition interaction on scores

19. Secondary Outcome: Trait Anxiety for Younger Adults
Description: Emotional well-being measured by the Trait Anxiety Inventory (TAI) for younger adults.
  The TAI consists of 20 items that are rated on a 4-point scale as follows: 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Scores range from 20 to 80, with higher scores indicating greater trait anxiety.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 55 | 49
score on a scale
  Time 1 | 42.473 (9.933) | 41.306 (12.582)
  Time 2 | 38.909 (9.487) | 38.510 (10.679)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.602, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores
Statistical Analysis 2: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.562, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 2]; p-value reflects effect of interest, a time x condition interaction on scores

20. Secondary Outcome: Trait Anxiety for Older Adults
Description: Emotional well-being measured by the Trait Anxiety Inventory (TAI) for older adults.
  The TAI consists of 20 items that are rated on a 4-point scale as follows: 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Scores range from 20 to 80, with higher scores indicating greater trait anxiety.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 28 | 27
score on a scale
  Time 1 | 33.821 (11.039) | 38.815 (12.830)
  Time 2 | 31.929 (9.071) | 36.093 (10.517)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.697, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores
Statistical Analysis 2: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.901, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 2]; p-value reflects effect of interest, a time x condition interaction on scores

21. Secondary Outcome: Stress Recovery (Systolic Blood Pressure) for Younger Adults
Description: Difference in stress recovery elicited by standard cognitive tasks, as assessed by change in systolic blood pressure from cognitive tasks to recovery rest
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 50 | 45
mmHg
  Time 1 | -2.993 (8.176) | -3.253 (6.465)
  Time 2 | -1.973 (6.728) | -0.702 (10.165)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.516, ANOVA; p-value reflects effect of interest, a time x condition interaction

22. Secondary Outcome: Stress Recovery (Systolic Blood Pressure) for Older Adults
Description: as for outcome 21
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 23 | 22
mmHg
  Time 1 | -6.464 (19.150) | -6.650 (6.060)
  Time 2 | -4.592 (17.651) | -4.380 (7.402)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.944, ANOVA; p-value reflects effect of interest, a time x condition interaction

23. Secondary Outcome: Stress Recovery (Heart Rate) for Younger Adults
Description: Difference in stress recovery elicited by standard cognitive tasks, as assessed by change in heart rate from cognitive tasks to recovery rest
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 31 | 30
beats per minute
  Time 1 | -3.851 (6.585) | -1.870 (4.133)
  Time 2 | -2.302 (4.658) | -1.486 (3.734)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.285, ANOVA; p-value reflects effect of interest, a time x condition interaction

24. Secondary Outcome: Stress Recovery (Heart Rate) for Older Adults
Description: as for outcome 23
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 13 | 16
beats per minute
  Time 1 | -3.921 (4.760) | -2.188 (2.111)
  Time 2 | -2.716 (2.921) | -1.267 (2.894)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.807, ANOVA; p-value reflects effect of interest, a time x condition interaction

25. Secondary Outcome: Stress Recovery (Breathing Rate) for Younger Adults
Description: Difference in stress recovery elicited by standard cognitive tasks, as assessed by change in breathing rate from cognitive tasks to recovery rest
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 46 | 40
breaths per minute
  Time 1 | -3.555 (3.121) | -4.134 (3.097)
  Time 2 | -4.722 (4.070) | -1.563 (2.533)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p < 0.001, ANOVA; p-value reflects effect of interest, a time x condition interaction

26. Secondary Outcome: Stress Recovery (Breathing Rate) for Older Adults
Description: as for outcome 25
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 18 | 18
breaths per minute
  Time 1 | -3.935 (2.487) | -3.194 (3.589)
  Time 2 | -4.046 (4.169) | -3.864 (4.262)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.740, ANOVA; p-value reflects effect of interest, a time x condition interaction

27. Secondary Outcome: Stress Reactivity (Systolic Blood Pressure) for Younger Adults
Description: Difference in stress reactivity elicited by standard cognitive tasks, as assessed by change in systolic blood pressure from rest to cognitive tasks
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 51 | 45
mmHg
  Time 1 | 3.090 (10.659) | 1.424 (8.867)
  Time 2 | -0.729 (8.402) | 1.812 (7.864)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.083, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores

28. Secondary Outcome: Stress Reactivity (Systolic Blood Pressure) for Older Adults
Description: as for outcome 27
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 23 | 23
mmHg
  Time 1 | 6.303 (12.349) | 6.196 (12.727)
  Time 2 | 6.553 (12.311) | 0.043 (11.351)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.176, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores

29. Secondary Outcome: Stress Reactivity (Heart Rate) for Younger Adults
Description: Difference in stress reactivity elicited by standard cognitive tasks, as assessed by change in heart rate from rest to cognitive tasks
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 32 | 29
beats per minute
  Time 1 | 4.270 (5.168) | 3.969 (5.085)
  Time 2 | 2.060 (3.776) | 2.951 (4.242)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.325, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores

30. Secondary Outcome: Stress Reactivity (Heart Rate) for Older Adults
Description: Difference in stress reactivity elicited by standard cognitive tasks, as assessed by change in heart rate from cognitive tasks to recovery rest
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 14 | 18
beats per minute
  Time 1 | 3.991 (3.987) | 3.555 (2.138)
  Time 2 | 2.731 (2.977) | 1.951 (3.099)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.751, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores

31. Secondary Outcome: Stress Reactivity (Breathing Rate) for Younger Adults
Description: Difference in stress reactivity elicited by standard cognitive tasks, as assessed by change in breathing rate from rest to cognitive tasks
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 47 | 38
breaths per minute
  Time 1 | 3.437 (3.096) | 3.367 (2.509)
  Time 2 | 4.381 (4.082) | 2.235 (2.023)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.011, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores

32. Secondary Outcome: Stress Reactivity (Breathing Rate) for Older Adults
Description: as for outcome 31
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 19 | 18
breaths per minute
  Time 1 | 4.287 (2.342) | 3.975 (3.986)
  Time 2 | 3.975 (4.122) | 3.895 (3.590)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.885, ANOVA; p-value reflects effect of interest, a time x condition interaction on scores

33. Secondary Outcome: Arterial Spin Labeling (ASL) for Younger Adults
Description: Cerebral blood flow was measured at pre-training resting state and post-training paced-breathing.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL/100 g/min
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 26 | 27
mL/100 g/min
  Time 1 | 44.01 (1.68) | 40.96 (1.53)
  Time 2 | 39.69 (1.61) | 38.98 (1.48)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; 2 (time) x 2 (condition) ANOVA to test effects of time, condition, and time x condition interaction; Test type: Superiority; p = 0.259, ANOVA — p-value reflects time x condition interaction

34. Secondary Outcome: Arterial Spin Labeling (ASL) for Older Adults
Description: Cerebral blood flow was measured at pre-training resting state and post-training paced-breathing.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL/100 g/min
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 13 | 17
mL/100 g/min
  Time 1 | 42.06 (2.33) | 40.86 (3.04)
  Time 2 | 30.95 (2.02) | 39.93 (1.89)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; 2 (time) x 2 (condition) ANOVA to test effects of time, condition, and time x condition interaction; Test type: Superiority; p = 0.000146, ANOVA — p-value reflects time x condition interaction

35. Secondary Outcome: High Frequency (HF) HRV for Younger Adults
Description: HRV measured by high frequency (HF) HRV for younger adults.
  HF-HRV was quantified as the spectral power of interbeat interval variability within the high frequency range (typically 0.15-0.40 Hz), which reflects parasympathetic (vagal) activity. In this study, HF-HRV was obtained using photoplethysmography (PPG) methods. During a standardized resting condition, the device continuously recorded interbeat intervals. These data were then processed via spectral analysis to calculate the power in the high frequency band. Measurements are expressed in units of milliseconds squared (ms²). Higher HF-HRV values indicate increased parasympathetic modulation and are generally associated with improved autonomic regulation and better cognitive performance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log transformed power(ms^2)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 56 | 46
log transformed power(ms^2)
  Time 1 | 6.94 (1.13) | 6.77 (0.76)
  Time 2 | 6.63 (1.01) | 6.62 (1.00)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.463, ANOVA — time point x group (2 way) interaction

36. Secondary Outcome: High Frequency (HF) HRV for Older Adults
Description: HRV measured by high frequency (HF) HRV for older adults.
  HF-HRV was quantified as the spectral power of interbeat interval variability within the high frequency range (typically 0.15-0.40 Hz), which reflects parasympathetic (vagal) activity. In this study, HF-HRV was obtained using photoplethysmography (PPG) methods. During a standardized resting condition, the device continuously recorded interbeat intervals. These data were then processed via spectral analysis to calculate the power in the high frequency band. Measurements are expressed in units of milliseconds squared (ms²). Higher HF-HRV values indicate increased parasympathetic modulation and are generally associated with improved autonomic regulation and better cognitive performance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log transformed power(ms^2)
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 25 | 28
log transformed power(ms^2)
  Time 1 | 5.56 (0.89) | 5.40 (1.08)
  Time 2 | 5.78 (1.04) | 5.63 (1.16)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.990, ANOVA — time point x group (2 way) interaction

37. Secondary Outcome: Low Frequency (LF) HRV for Younger Adults
Description: HRV measured by low frequency (LF) HRV for younger adults.
  LF-HRV was quantified as the spectral power of interbeat interval variability within the low frequency range (typically 0.04-0.15 Hz), which reflects the combined influences of sympathetic and parasympathetic activity. In this study, LF-HRV was obtained using photoplethysmography (PPG) methods. During a standardized resting condition, the device continuously recorded interbeat intervals. These data were then processed via spectral analysis to calculate the power in the low frequency band. Measurements are expressed in units of milliseconds squared (ms²). Although LF-HRV reflects contributions from both branches of the autonomic nervous system, higher LF-HRV values can indicate enhanced autonomic modulation, with interpretation made in the context of overall autonomic balance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log transformed power(ms^2)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 56 | 46
log transformed power(ms^2)
  Time 1 | 7.25 (1.03) | 6.95 (0.93)
  Time 2 | 7.61 (1.21) | 6.75 (1.01)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.034, ANOVA — time point x group (2 way) interaction

38. Secondary Outcome: Low Frequency (LF) HRV for Older Adults
Description: HRV measured by low frequency (LF) HRV for older adults.
  LF-HRV was quantified as the spectral power of interbeat interval variability within the low frequency range (typically 0.04-0.15 Hz), which reflects the combined influences of sympathetic and parasympathetic activity. In this study, LF-HRV was obtained using photoplethysmography (PPG) methods. During a standardized resting condition, the device continuously recorded interbeat intervals. These data were then processed via spectral analysis to calculate the power in the low frequency band. Measurements are expressed in units of milliseconds squared (ms²). Although LF-HRV reflects contributions from both branches of the autonomic nervous system, higher LF-HRV values can indicate enhanced autonomic modulation, with interpretation made in the context of overall autonomic balance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log transformed power(ms^2)
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 25 | 28
log transformed power(ms^2)
  Time 1 | 5.66 (1.19) | 5.14 (1.39)
  Time 2 | 6.11 (1.49) | 5.31 (1.65)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.398, ANOVA — time point x group (2 way) interaction

39. Secondary Outcome: The Root Mean Squared Successive Differences (RMSSD) HRV for Younger Adults
Description: HRV measured by the root mean square of successive differences (RMSSD) for younger adults.
  RMSSD (Root Mean Square of Successive Differences) is a time-domain measure that quantifies the variability between successive interbeat intervals, primarily reflecting parasympathetic (vagal) activity. In this study, RMSSD was obtained using photoplethysmography (PPG) methods. During a standardized resting condition, the device continuously recorded interbeat intervals, and RMSSD was computed as the square root of the mean of the squared differences between consecutive interbeat intervals. Measurements are expressed in milliseconds (ms). Higher RMSSD values indicate increased parasympathetic modulation, generally associated with improved autonomic regulation and better cardiovascular and cognitive performance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 56 | 46
millisecond
  Time 1 | 68.99 (40.74) | 56.78 (20.81)
  Time 2 | 60.99 (28.36) | 61.78 (42.66)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.113, ANOVA — time point x group (2 way) interaction

40. Secondary Outcome: The Root Mean Squared Successive Differences (RMSSD) HRV for Older Adults
Description: HRV measured by the root mean square of successive differences (RMSSD) for older adults.
  RMSSD (Root Mean Square of Successive Differences) is a time-domain measure that quantifies the variability between successive interbeat intervals, primarily reflecting parasympathetic (vagal) activity. In this study, RMSSD was obtained using photoplethysmography (PPG) methods. During a standardized resting condition, the device continuously recorded interbeat intervals, and RMSSD was computed as the square root of the mean of the squared differences between consecutive interbeat intervals. Measurements are expressed in milliseconds (ms). Higher RMSSD values indicate increased parasympathetic modulation, generally associated with improved autonomic regulation and better cardiovascular and cognitive performance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 25 | 28
millisecond
  Time 1 | 33.99 (16.87) | 33.39 (15.07)
  Time 2 | 42.17 (26.05) | 39.09 (20.55)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.637, ANOVA — time point x group (2 way) interaction

41. Secondary Outcome: Inflammation Measured by C-reactive Protein for Younger Adults
Description: Inflammation measured by salivary C-reactive protein (CRP) for younger adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: CRP level (pg/ml)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 52 | 47
CRP level (pg/ml)
  Time 1 | 8193.259 (3905.210) | 4069.873 (4107.658)
  Time 2 | 6093.377 (3115.766) | 3985.363 (3277.311)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority — time x condition interaction in CRP for younger adults; p = 0.133, ANOVA

42. Secondary Outcome: Inflammation Measured by C-reactive Protein for Older Adults
Description: Inflammation measured by salivary C-reactive protein (CRP) for older adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: CRP level (pg/ml)
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 14 | 14
CRP level (pg/ml)
  Time 1 | 2809.771 (1063.422) | 864.984 (1063.422)
  Time 2 | 1440.859 (437.418) | 509.761 (437.418)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority — time x condition interaction in CRP for older adults; p = 0.402, ANOVA

43. Secondary Outcome: Inflammation Measured by IL-1b Levels for Younger Adults
Description: Inflammation measured by salivary IL-1b levels for younger adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IL-1b level (pg/ml)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 53 | 46
IL-1b level (pg/ml)
  Time 1 | 80.063 (15.825) | 91.827 (16.987)
  Time 2 | 86.474 (13.624) | 76.446 (14.624)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine IL-1b for younger adults; p = 0.236, ANOVA — p value for time x condition interaction effect

44. Secondary Outcome: Inflammation Measured by IL-1b Levels for Older Adults
Description: Inflammation measured by salivary IL-1b levels for older adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IL-1b level (pg/ml)
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 15 | 12
IL-1b level (pg/ml)
  Time 1 | 218.580 (73.483) | 89.007 (82.157)
  Time 2 | 174.882 (44.839) | 90.668 (50.131)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine IL-1b for older adults; p = 0.600, ANOVA — p value for time x condition interaction effect

45. Secondary Outcome: Inflammation Measured by IL-6 Levels for Younger Adults
Description: Inflammation measured by salivary IL-6 levels for younger adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IL-6 level (pg/ml)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 53 | 46
IL-6 level (pg/ml)
  Time 1 | 4.653 (0.858) | 3.571 (0.921)
  Time 2 | 4.510 (0.884) | 3.029 (0.949)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine IL-6 for younger adults; p = 0.788, ANOVA — p value for time x condition interaction effect

46. Secondary Outcome: Inflammation Measured by IL-6 Levels for Older Adults
Description: Inflammation measured by salivary IL-6 levels for older adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IL-6 level (pg/ml)
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 15 | 12
IL-6 level (pg/ml)
  Time 1 | 10.559 (4.439) | 7.595 (4.963)
  Time 2 | 8.260 (2.108) | 4.605 (2.357)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine IL-6 for older adults; p = 0.917, ANOVA — p value for time x condition interaction effect

47. Secondary Outcome: Inflammation Measured by IL-8 Levels for Younger Adults
Description: Inflammation measured by salivary IL-8 levels for younger adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IL-8 level (pg/ml)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 53 | 46
IL-8 level (pg/ml)
  Time 1 | 513.510 (89.567) | 540.543 (96.140)
  Time 2 | 448.990 (60.839) | 502.338 (65.304)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine IL-8 for younger adults; p = 0.844, ANOVA — p value for time x condition interaction effect

48. Secondary Outcome: Inflammation Measured by IL-8 Levels for Older Adults
Description: Inflammation measured by salivary IL-8 levels for older adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IL-8 level (pg/ml)
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 15 | 12
IL-8 level (pg/ml)
  Time 1 | 1440.907 (270.644) | 656.653 (302.589)
  Time 2 | 1343.894 (273.858) | 698.642 (306.182)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine IL-8 for older adults; p = 0.750, ANOVA — p value for time x condition interaction effect

49. Secondary Outcome: Inflammation Measured by TNF-a Levels for Younger Adults
Description: Inflammation measured by salivary TNF-a levels for younger adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: TNF-a level (pg/ml)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 53 | 46
TNF-a level (pg/ml)
  Time 1 | 2.792 (0.367) | 2.947 (0.394)
  Time 2 | 3.241 (0.411) | 2.202 (0.441)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine TNF-a for younger adults; p = 0.074, ANOVA — p value for time x condition interaction effect

50. Secondary Outcome: Inflammation Measured by TNF-a Levels for Older Adults
Description: Inflammation measured by salivary TNF-a levels for older adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: TNF-a level (pg/ml)
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 15 | 12
TNF-a level (pg/ml)
  Time 1 | 4.271 (0.945) | 1.607 (1.056)
  Time 2 | 3.887 (0.985) | 2.338 (1.101)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority — time x condition interaction in cytokine TNF-a for older adults; p = 0.0505, ANOVA — p value for time x condition interaction effect

51. Secondary Outcome: Plasma Amyloid Beta 40 (Aβ40) for Younger Adults
Description: Plasma Aβ40 levels at pre- and post-intervention were compared between HRV-increase and HRV-decrease group for younger adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 30 | 24
pg/ml
  Time 1 (pre-intervention) | 166.95 (7.58) | 151.75 (4.95)
  Time 2 (post-intervention) | 150.25 (7.16) | 172.16 (7.87)

52. Secondary Outcome: Plasma Amyloid Beta 40 (Aβ40) for Older Adults
Description: Plasma Aβ40 levels at pre- and post-intervention were compared between HRV-increase and HRV-decrease group for older adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 27 | 27
pg/ml
  Time 1 (pre-intervention) | 198.02 (9.15) | 211.76 (23.47)
  Time 2 (post-intervention) | 189.95 (12.76) | 227.99 (19.85)

53. Secondary Outcome: Plasma Amyloid Beta 42 (Aβ42) Younger Adults
Description: Plasma Aβ42 levels at pre- and post-intervention were compared between HRV-increase and HRV-decrease group for younger adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 30 | 24
pg/ml
  Time 1 (pre-intervention) | 9.77 (0.43) | 9.26 (0.47)
  Time 2 (post-intervention) | 8.85 (0.46) | 10.84 (0.74)

54. Secondary Outcome: Plasma Amyloid Beta 42 (Aβ42) for Older Adults
Description: Plasma Aβ42 levels at pre- and post-intervention were compared between HRV-increase and HRV-decrease group for older adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 27 | 27
pg/ml
  Time 1 (pre-intervention) | 10.78 (0.58) | 10.54 (0.75)
  Time 2 (post-intervention) | 10.94 (0.62) | 11.80 (0.55)

55. Secondary Outcome: Plasma Phosphorylated Tau 181 (pTau) for Younger Adults
Description: Plasma pTau levels at pre- and post-intervention were reported for HRV-increase and HRV-decrease group for younger adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 30 | 24
pg/ml
  Time 1 (pre-intervention) | 1.57 (0.12) | 1.57 (0.14)
  Time 2 (post-intervention) | 1.63 (0.12) | 1.66 (0.15)

56. Secondary Outcome: Plasma Phosphorylated Tau 181 (pTau) for Older Adults
Description: Plasma pTau levels at pre- and post-intervention were compared between HRV-increase and HRV-decrease group for older adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 27 | 27
pg/ml
  Time 1 (pre-intervention) | 2.55 (0.22) | 2.94 (0.36)
  Time 2 (post-intervention) | 2.64 (0.31) | 2.29 (0.26)

57. Secondary Outcome: Plasma Total Tau (tTau) for Younger Adults
Description: Plasma tTau levels at pre- and post-intervention were reported for HRV-increase and HRV-decrease group for younger adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 30 | 24
pg/ml
  Time 1 (pre-intervention) | 2.13 (0.14) | 2.11 (0.16)
  Time 2 (post-intervention) | 1.87 (0.12) | 2.55 (0.20)

58. Secondary Outcome: Plasma Total Tau (tTau) for Older Adults
Description: Plasma tTau levels at pre- and post-intervention were compared between HRV-increase and HRV-decrease group for older adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 27 | 27
pg/ml
  Time 1 (pre-intervention) | 1.91 (0.12) | 2.07 (0.17)
  Time 2 (post-intervention) | 2.17 (0.22) | 2.13 (0.12)

59. Secondary Outcome: LC-innervated Subregion Volume in the Hippocampus for Younger Adults
Description: LC-innervated subregion volume in the hippocampus at pre- and post-intervention was compared between the HRV-increase and HRV-decrease groups in younger adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 49 | 47
mm^3
  Time 1 (pre-intervention) | 1177.99 (15.00) | 1142.29 (15.32)
  Time 2 (post-intervention) | 1172.27 (15.01) | 1142.45 (15.33)

60. Secondary Outcome: LC-innervated Subregion Volume in the Hippocampus for Older Adults
Description: LC-innervated subregion volume in the hippocampus at pre- and post-intervention was compared between the HRV-increase and HRV-decrease groups in older adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 23 | 25
mm^3
  Time 1 (pre-intervention) | 1095.66 (23.58) | 1126.17 (22.62)
  Time 2 (post-intervention) | 1106.20 (24.18) | 1110.82 (22.62)

61. Secondary Outcome: Cortical Volume in the Left Orbitofrontal Cortex for Younger Adults
Description: Left orbitofrontal volume at pre- and post-intervention was compared between the HRV-increase and HRV-decrease groups in younger adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 49 | 47
mm^3
  Time 1 (pre-intervention) | 14001.81 (119.80) | 14024.90 (122.34)
  Time 2 (post-intervention) | 14055.29 (125.81) | 13878.29 (128.47)

62. Secondary Outcome: Cortical Volume in the Left Orbitofrontal Cortex for Older Adults
Description: Left orbitofrontal volume at pre- and post-intervention was compared between the HRV-increase and HRV-decrease groups in older adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 23 | 25
mm^3
  Time 1 (pre-intervention) | 12369.59 (146.40) | 12391.75 (143.44)
  Time 2 (post-intervention) | 12452.50 (152.74) | 12290.84 (149.65)

63. Secondary Outcome: Cortical Volume in the Right Orbitofrontal Cortex for Younger Adults
Description: Right orbitofrontal volume at pre- and post-intervention was compared between the HRV-increase and HRV-decrease groups in younger adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 49 | 47
mm^3
  Time 1 (pre-intervention) | 14231.64 (132.05) | 14005.03 (134.84)
  Time 2 (post-intervention) | 14233.22 (132.08) | 13898.56 (134.87)

64. Secondary Outcome: Cortical Volume in the Right Orbitofrontal Cortex for Older Adults
Description: Right orbitofrontal volume at pre- and post-intervention was compared between the HRV-increase and HRV-decrease groups in older adults.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 23 | 25
mm^3
  Time 1 (pre-intervention) | 12246.75 (150.82) | 12582.37 (147.77)
  Time 2 (post-intervention) | 12278.02 (157.55) | 12540.15 (154.36)

65. Secondary Outcome: mPFC-left Amygdala Resting-state Functional Connectivity for Younger Adults (Post-Pre)
Description: The strength of resting-state functional connectivity between mPFC and the left amygdala was measured by correlation coefficients. The difference in functional connectivity between the two time points (Time 2 - Time 1) was calculated. Higher values indicate greater connectivity at Time 2 than Time 1 (or post- than pre-intervention).
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 49 | 47
correlation coefficients | 0.093 (0.040) | -0.018 (0.025)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; An independent t-test was performed to compare the two groups; Test type: Superiority; p = 0.022, t-test, 2 sided

66. Secondary Outcome: mPFC-left Amygdala Resting-state Functional Connectivity for Older Adults (Post-Pre)
Description: as for outcome 65
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 26 | 25
correlation coefficients | 0.002 (0.080) | 0.074 (0.051)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; An independent t-test was performed to compare the two groups; Test type: Superiority; p = 0.455, t-test, 2 sided

67. Secondary Outcome: mPFC-left Amygdala Resting-state Functional Connectivity for Younger Adults (ANOVA)
Description: The strength of resting-state functional connectivity was measured by correlation coefficients. Values represent the correlation of BOLD time-series between mPFC and the left amygdala. Higher values indicate greater connectivity.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 49 | 47
correlation coefficients
  Time 1 | 0.076 (0.021) | 0.089 (0.022)
  Time 2 | 0.168 (0.021) | 0.072 (0.021)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; A 2 (time: pre, post) X 2 (condition: HRV-increase, HRV-decrease) ANOVA was performed; Test type: Superiority; p = 0.022, ANOVA

68. Secondary Outcome: mPFC-left Amygdala Resting-state Functional Connectivity for Older Adults (ANOVA)
Description: as for outcome 67
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correlation coefficients
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 26 | 25
correlation coefficients
  Time 1 | 0.200 (0.050) | 0.079 (0.051)
  Time 2 | 0.202 (0.048) | 0.153 (0.049)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; A 2 (time: pre, post) X 2 (condition: HRV-increase, HRV-decrease) ANOVA was performed; Test type: Superiority; p = 0.455, ANOVA

69. Other Pre Specified Outcome: Working Memory for Younger Adults
Description: Working memory performance measured by NIH Toolbox List Sorting Working Memory Test (LSWM). The standard score is calculated to have a normative mean of 100 and a standard deviation (SD) of 15. Scores range from 59 to 140, with higher scores indicating better Working memory.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: age corrected standard score
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 56 | 49
age corrected standard score
  Time 1 | 98.39 (10.35) | 98.04 (14.00)
  Time 2 | 105.13 (10.39) | 103.10 (12.21)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.462, ANOVA — time point x group (2 way) interaction

70. Other Pre Specified Outcome: Working Memory for Older Adults
Description: as for outcome 69
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: age corrected standard score
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 31 | 28
age corrected standard score
  Time 1 | 102.48 (14.82) | 101.29 (14.14)
  Time 2 | 103.06 (13.95) | 104.82 (11.16)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.305, ANOVA — time point x group (2 way) interaction

71. Other Pre Specified Outcome: Processing Speed for Younger Adults
Description: Processing speed performance measured by NIH Toolbox Pattern Comparison Processing Speed Test (PCPS).
  The standard score is calculated to have a normative mean of 100 and a standard deviation (SD) of 15. Scores range from 59 to 140, with higher scores indicating faster processing speed.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: age corrected standard score
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 56 | 49
age corrected standard score
  Time 1 | 102.64 (22.69) | 105.55 (18.53)
  Time 2 | 116.30 (17.72) | 118.51 (16.08)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.804, ANOVA — time point x group (2 way) interaction

72. Other Pre Specified Outcome: Processing Speed for Older Adults
Description: as for outcome 71
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: age corrected standard score
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 31 | 28
age corrected standard score
  Time 1 | 106.55 (21.10) | 98.54 (20.96)
  Time 2 | 107.68 (25.53) | 105.43 (17.57)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.141, ANOVA — time point x group (2 way) interaction

73. Other Pre Specified Outcome: Inhibitory Control and Attention for Younger Adults
Description: Inhibitory control performance measured by NIH Toolbox Flanker Inhibitory Control and Attention Test (Flanker).
  The standard score is calculated to have a normative mean of 100 and a standard deviation (SD) of 15. Scores range from 59 to 140, with higher scores indicating better Inhibitory Control and Attention.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: age corrected standard score
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 56 | 49
age corrected standard score
  Time 1 | 87.27 (14.29) | 84.90 (12.17)
  Time 2 | 89.21 (15.03) | 88.71 (11.96)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Test type: Superiority; p = 0.292, ANOVA — time point x group(2 way) interaction

74. Other Pre Specified Outcome: Inhibitory Control and Attention for Older Adults
Description: as for outcome 73
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: age corrected standard score
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 31 | 28
age corrected standard score
  Time 1 | 90.84 (8.91) | 89.82 (11.17)
  Time 2 | 93.29 (8.76) | 92.04 (13.44)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Test type: Superiority; p = 0.905, ANOVA — time point x group (2 way) interaction

75. Other Pre Specified Outcome: Sustained Attention for Younger Adults
Description: Sustained attention performance was measured by Sustained Attention to Response Test (SART).
  A commission error was calculated as the number of button press for 25 no-go trials, and an omission error was calculated as the number of no button press for 200 go trials in younger adults. The number of errors range from 0 to 25 for commission errors and from 0 to 200 for omission errors. A higher number of omission and commission errors indicates worse sustained attention performance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number of errors
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 53 | 47
number of errors
  Time 1: commission error | 12.679 (0.936) | 12.979 (0.994)
  Time 2: commission error | 9.830 (1.041) | 9.851 (1.106)
  Time 1: omission error | 1.906 (0.592) | 3.383 (0.628)
  Time 2: omission error | 1.792 (0.541) | 2.383 (0.574)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; time x condition x error type interaction in Sustained Attention to Response Task (SART) for younger adults; Test type: Superiority; p = 0.641, ANOVA — p value for time x condition x error type interaction effect

76. Other Pre Specified Outcome: Sustained Attention for Older Adults
Description: Sustained attention performance was measured by Sustained Attention to Response Test (SART).
  A commission error was calculated as the number of button press for 25 no-go trials, and an omission error was calculated as the number of no button press for 200 go trials in older adults. The number of errors range from 0 to 25 for commission errors and from 0 to 200 for omission errors. A higher number of omission and commission errors indicates worse sustained attention performance.
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number of errors
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 26 | 19
number of errors
  Time 1: commission error | 9.538 (1.172) | 9.211 (1.371)
  Time 2: commission error | 8.692 (1.152) | 8.789 (1.347)
  Time 1: omission error | 3.731 (1.187) | 4.947 (1.389)
  Time 2: omission error | 1.731 (0.765) | 2.842 (0.894)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; time x condition x error type interaction in Sustained Attention to Response Task (SART) for older adults; Test type: Superiority; p = 0.813, ANOVA — p value for time x condition x error type interaction effect

77. Other Pre Specified Outcome: Recognition Memory for Younger Adults (Hits)
Description: Recognition memory performance based on average proportion of previously presented images that were correctly identified (i.e., hits) by younger adults
Time Frame: Week 5 Lab Visit (after about 2.5-3 weeks of training)
Population: Population analyzed was composed by all randomization subjects who completed the memory tests and whose data quality was sufficient for data analysis.
Measure: Mean (Standard Error); unit: Proportion of correct hits
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 55 | 50
Proportion of correct hits
  Neutral | .880 (.014) | .873 (.013)
  Positive | .886 (.012) | .866 (.011)
  Negative | .914 (.011) | .900 (.012)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Hits during recognition task for younger adults; Test type: Superiority; p = .695, ANOVA

78. Other Pre Specified Outcome: Recognition Memory for Older Adults (Hits)
Description: Recognition memory performance based on average proportion of previously presented images that were correctly identified (i.e., hits) by older adults
Time Frame: Week 5 Lab Visit (after about 2.5-3 weeks of training)
Population: as for outcome 77
Measure: Mean (Standard Error); unit: Proportion of correct hits
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 29 | 31
Proportion of correct hits
  Neutral | .828 (.020) | .859 (.015)
  Positive | .820 (.022) | .851 (.016)
  Negative | .875 (.017) | .870 (.014)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Hits during recognition task for older adults; Test type: Superiority; p = .270, ANOVA

79. Other Pre Specified Outcome: Recognition Memory for Younger Adults (False Alarm)
Description: Recognition memory performance based on average proportion of images not previously presented that were incorrectly identified as seen (i.e., False Alarms) by younger adults
Time Frame: Week 5 Lab Visit (after about 2.5-3 weeks of training)
Population: as for outcome 77
Measure: Mean (Standard Error); unit: Proportion of false alarm
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 55 | 50
Proportion of false alarm
  Neutral | .048 (.007) | .042 (.006)
  Positive | .044 (.008) | .046 (.008)
  Negative | .027 (.005) | .041 (.007)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; False alarms during recognition task for younger adults; Test type: Superiority; p = .102, ANOVA

80. Other Pre Specified Outcome: Recognition Memory for Older Adults (False Alarm)
Description: Recognition memory performance based on average proportion of images not previously presented that were incorrectly identified as seen (i.e., False Alarms) by older adults
Time Frame: Week 5 Lab Visit (after about 2.5-3 weeks of training)
Population: as for outcome 77
Measure: Mean (Standard Error); unit: Proportion of false alarms
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 29 | 31
Proportion of false alarms
  Neutral | .091 (.017) | .047 (.011)
  Positive | .093 (.018) | .062 (.011)
  Negative | .069 (.012) | .052 (.011)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; False alarms during recognition task for older adults; Test type: Superiority; p = .257, ANOVA

81. Other Pre Specified Outcome: Recall Memory for Younger Adults
Description: Average proportion of previously presented images that were correctly recalled by younger adults
Time Frame: Week 5 Lab Visit (after about 2.5-3 weeks of training)
Population: as for outcome 77
Measure: Mean (Standard Error); unit: Proportion of items correctly recalled
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 52 | 50
Proportion of items correctly recalled
  Positive | .285 (.023) | .214 (.023)
  Negative | .248 (.020) | .262 (.027)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; Group difference for recall for younger adults; Test type: Superiority; p = .067, ANOVA

82. Other Pre Specified Outcome: Recall Memory for Older Adults
Description: Average proportion of previously presented images that were correctly recalled by older adults
Time Frame: Week 5 Lab Visit (after about 2.5-3 weeks of training)
Population: as for outcome 77
Measure: Mean (Standard Error); unit: Proportion of items correctly recalled
Arm/Group | Older HRV-increase Group | Older HRV-decrease Group
Number analyzed (Participants) | 27 | 28
Proportion of items correctly recalled
  Positive | .203 (.030) | .156 (.025)
  Negative | .225 (.036) | .286 (.040)
Statistical Analysis 1: Comparison: Older HRV-increase Group vs Older HRV-decrease Group; Group difference for recall for older adults; Test type: Superiority; p = .117, ANOVA

83. Other Pre Specified Outcome: Stress Measured by Cortisol Levels for Younger Adults
Description: Stress measured by salivary cortisol levels for younger adults
Time Frame: Time 1 (Baseline), Time 2 (5 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: CAR level (µg/dL)
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group
Number analyzed (Participants) | 50 | 44
CAR level (µg/dL)
  Time 1: cortisol level at awakening | 0.231 (0.023) | 0.248 (0.024)
  Time 1: cortisol level at 30 min after awakening | 0.431 (0.035) | 0.453 (0.037)
  Time 2: cortisol level at awakening | 0.284 (0.033) | 0.309 (0.035)
  Time 2: cortisol level at 30 min after awakening | 0.478 (0.045) | 0.472 (0.048)
Statistical Analysis 1: Comparison: Younger HRV-increase Group vs Younger HRV-decrease Group; time x condition x collection interaction in cortisol levels for younger adults; Test type: Superiority; p = 0.558, ANOVA — p value for time x condition interaction effect

ADVERSE EVENTS:
Time Frame: 7 weeks
Groups:
- Younger HRV-increase Group: Participants in this group are between the ages of 18 and 35.
  Half of the younger participants will be randomly assigned to this group who will undergo daily practice to increase their heart rate variability (HRV).
- Younger HRV-decrease Group: Participants in this group are between the ages of 18 and 35.
  Half of the younger participants will be randomly assigned to this group who will undergo daily practice to decrease their heart rate variability (HRV).
- Older HRV-increase Group: Participants in this group are between the ages of 55 and 80.
  Half of the older participants will be randomly assigned to this group who will undergo daily practice to increase their heart rate variability (HRV).
- Older HRV-decrease Group: Participants in this group are between the ages of 55 and 80.
  Half of the older participants will be randomly assigned to this group who will undergo daily practice to decrease their heart rate variability (HRV).
Arm/Group | Younger HRV-increase Group | Younger HRV-decrease Group | Older HRV-increase Group | Older HRV-decrease Group
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/58 | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/58 | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 0/63 | 0/58 | 0/37 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT03458910/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT03458910/SAP_001.pdf